CLINICAL TRIAL: NCT04281472
Title: A Phase 2 Trial to Investigate the Efficacy, Safety, and Tolerability of Efgartigimod PH20 SC in Adult Patients With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: A Study to Assess the Safety and Efficacy of a Subcutaneous Formulation of Efgartigimod in Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP, an Autoimmune Disorder That Affects the Peripheral Nerves)
Acronym: ADHERE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1802; 2019-003076-39 (EudraCT Number)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- efgartigimod PH20 SC (Experimental): patients receiving efgartigimod PH20 SC in both stage A as stage B
  Interventions: Biological: efgartigimod PH20 SC in stage B
- Placebo (Placebo Comparator): patients receiving efgartigimod PH20 SC during stage A and receiving placebo in stage B
  Interventions: Biological: efgartigimod PH20 SC in stage B; Other: placebo in stage B

INTERVENTIONS:
Biological: efgartigimod PH20 SC in stage B — Stage A: efgartigimod PH20 SC, Stage B: efgartigimod PH20 SC
Other: placebo in stage B — Stage A: N/A, stage B: placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2 study to evaluate the safety and efficacy of the subcutaneous formulation of efgartigimod in adults with CIDP.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the requirements of the trial, provide written informed consent (include consent for the use and disclosure of research-related health information), willingness and ability to comply with the trial protocol procedures (including required trial visits)
2. Male or female patient aged 18 years or older, at the time of signing the informed consent.
3. Diagnosed with probable or definite CIDP according to criteria of the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS 2010), progressing or relapsing forms.
4. CIDP Disease Activity Status (CDAS) score ≥2 at screening.
5. INCAT score ≥2 at the first run-in visit (for patients entering run-in) or stage A baseline (for treatment-naïve patients with documented evidence for worsening on the total adjusted INCAT disability score within 3 months prior to screening). Patients with an INCAT score of 2 at trial entry must have this score exclusively from the leg disability score; for patients with an INCAT score of ≥3 at trial entry, there are no specific requirements for arm or leg scores.
6. Fulfilling any of the following treatment conditions:

   * Currently treated with pulsed corticosteroids, oral corticosteroids equivalent to prednisolone/prednisone ≤10mg/day, and/or IVIg or SCIg, if this treatment has been started within the last 5 years before screening, and the patient is willing to discontinue this treatment at the first run-in visit; or
   * Without previous treatment (treatment-naive); or
   * Treatment with corticosteroids and/or IVIg or SCIg discontinued at least 6 months prior to screening Note: Patients not treated with monthly or daily corticosteroids, IVIg or SCIg for at least 6 months prior to screening are considered as equal to treatment-naïve patients.
7. Women of childbearing potential who have a negative pregnancy test at screening and a negative urine pregnancy test up to Stage A baseline.
8. Women of childbearing potential must use an acceptable method of contraception from signing the ICF until the date of the last dose of IMP

Exclusion Criteria:

1. Pure sensory atypical CIDP (EFNS/PNS definition).
2. Polyneuropathy of other causes, including the following: Multifocal motor neuropathy; Monoclonal gammopathy of uncertain significance with anti-myelin associated, glycoprotein immunoglobulin M (IgM) antibodies; Hereditary demyelinating neuropathy; Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin change syndromes; Lumbosacral radiculoplexus neuropathy; Polyneuropathy most likely due to diabetes mellitus; Polyneuropathy most likely due to systemic illnesses; Drug- or toxin-induced polyneuropathy.
3. Any other disease that could better explain the patient's signs and symptoms.
4. Any history of myelopathy or evidence of central demyelination.
5. Current or past history (within 12 months of screening) of alcohol, drug or medication abuse.
6. Severe psychiatric disorder (such as severe depression, psychosis, bipolar disorder), history of suicide attempt, or current suicidal ideation that in the opinion of the investigator could create undue risk to the patient or could affect adherence with the trial protocol.
7. Patients with clinically significant active or chronic uncontrolled bacterial, viral, or fungal infection at screening, including patients who test positive for an active viral infection at screening with: Active Hepatitis B Virus (HBV): serologic panel test results indicative of an active (acute or chronic) infection; Active Hepatitis C Virus (HCV): serology positive for HCV-Ab; Human Immunodeficiency Virus (HIV) positive serology associated with an Acquired Immune Deficiency Syndrome (AIDS)-defining condition or with a cluster of differentiation 4 (CD4) count ≤200 cells/mm3.
8. Total IgG level <6 g/L at screening.
9. Treatment with the following: Within 3 months (or 5 half-lives of the drug, whichever is longer) before screening: plasma exchange or immunoadsorption, any concomitant Fc-containing therapeutic agents or other biological, or any other investigational product; Within 6 months before screening: rituximab, alemtuzumab, any other monoclonal antibody, cyclophosphamide, interferon, tumor necrosis factor-alpha inhibitors, fingolimod, methotrexate, azathioprine, mycophenolate, any other immunomodulating or immunosuppressive medications, and oral daily corticosteroids >10 mg/day. Note: Patients using IVIg, SCIg, pulsed corticosteroids, and oral daily corticosteroids ≤10 mg/day can be included.

   Patients who (intend to) use prohibited medications and therapies (see protocol) during the trial.
10. Pregnant and lactating women and those intending to become pregnant during the trial or within 90 days after last IMP administration.
11. Patients with any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of CIDP.
12. Patients who received a live-attenuated vaccine fewer than 28 days before screening. Receiving an inactivated, sub-unit, polysaccharide, or conjugate vaccine any time before screening is not exclusionary.
13. Patients who have a history of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before the first IMP administration. Patients with the following cancer can be included anytime: Adequately treated basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, or Incidental histological finding of Prostate cancer (TNM [tumor, nodes, and metastases classification] stage T1a or T1b).
14. Patients who previously participated in a trial with efgartigimod and have received at least one administration of IMP.
15. Patients with known medical history of hypersensitivity to any of the ingredients of IMP.
16. Patients with clinical evidence of other significant serious disease or patients who underwent a recent or have a planned major surgery, or any other reason which could confound the results of the trial or put the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (215):
- United States (45):
  - Investigator site 0010065, Birmingham, Alabama
  - Investigator site 0010013, Phoenix, Arizona
  - Investigator site 0010055, Scottsdale, Arizona
  - Investigator Site 0010032, Carlsbad, California
  - Investigator site 0010004, Orange, California
  - Investigator site 0010190, Pomona, California
  - Investigator site 0010160, Rancho Mirage, California
  - Investigator site 0010071, San Francisco, California
  - Investigator site 0010057, Centennial, Colorado
  - Investigator site 0010026, New Haven, Connecticut
  - Investigator site 0010072, Boca Raton, Florida
  - Investigator site 0010144, Coral Springs, Florida
  - Investigator site 0010023, Jacksonville, Florida
  - Investigator Site 0010068, Maitland, Florida
  - Investigator site 0010059, Miami, Florida
  - Investigator site 0010050, Orlando, Florida
  - Investigator site 0010172, Ormond Beach, Florida
  - Investigator site 0010006, Tampa, Florida
  - Investigator site 0010125, Augusta, Georgia
  - Investigator site 0010011, Iowa City, Iowa
  - Investigator site 0010015, Fairway, Kansas
  - Investigator site 0010147, Lexington, Kentucky
  - Investigator site 0010014, Detroit, Michigan
  - Investigator site 0010063, East Lansing, Michigan
  - Investigator site 0010052, Minneapolis, Minnesota
  - Investigator site 0010028, Columbia, Missouri
  - Investigator site 0010070, New Brunswick, New Jersey
  - Investigator site 0010069, New York, New York
  - Investigator site 0010168, New York, New York
  - Investigator site 0010191, New York, New York
  - Investigator site 0010074, New York, New York
  - Investigator site 0010075, Patchogue, New York
  - Investigator site 0010003, Chapel Hill, North Carolina
  - Investigator site 0010077, Durham, North Carolina
  - Investigator site 0010051, Cincinnati, Ohio
  - Investigator site 0010064, Columbus, Ohio
  - Investigator site 0010047, Philadelphia, Pennsylvania
  - Investigator site 0010007, Philadelphia, Pennsylvania
  - Investigator site 0010067, Pittsburgh, Pennsylvania
  - Investigator site 0010066, Austin, Texas
  - Investigator site 0010026, Houston, Texas
  - Investigator site 0010009, San Antonio, Texas
  - Investigator site 0010076, Burlington, Vermont
  - Investigator site 0010007, Charlottesville, Virginia
  - Investigator site 0010061, Richmond, Virginia
- Austria (5):
  - Investigator site 0430009, Graz
  - Investigator site 0430007, Innsbruck
  - Investigator site 0430008, Linz
  - Investigator site 0430006, Salzburg
  - Investigator site 0430005, Vienna
- Belgium (6):
  - Investigator site 0320017, Brussels
  - Investigator site 0320019, Brussels
  - Investigator site 0320016, Edegem
  - Investigator site 0320009, Leuven
  - Investigator site 0320024, Liège
  - Investigator site 0320022, Woluwe-Saint-Lambert
- Bulgaria (4):
  - Investigator site 3590007, Pleven
  - Investigator site 3590008, Sofia
  - Investigator site 3590009, Sofia
  - Investigator site 3590005, Sofia
- China (26):
  - Investigator site 0860033, Beijing
  - Investigator site 0860030, Changchun
  - Investigator site 0860041, Changsha
  - Investigator site 0860036, Chengdu
  - Investigator site 0860049, Chifeng
  - Investigator site 0860038, Fuzhou
  - Investigator site 0860050, Guanzhou
  - Investigator site 0860032, Guanzhou
  - Investigator site 0860045, Guiyang
  - Investigator site 0860046, Hangzhou
  - Investigator site 0860035, Hanzhou
  - Investigator site 0860031, Jinan
  - Investigator site 0860063, Jining
  - Investigator site 0860044, Nanchang
  - Investigator Site 0860040, Nanchang
  - Investigator site 0860051, Nanchang
  - Investigator site 0860043, Nanjing
  - Investigator site 0860047, Shanghai
  - Investigator site 0860028, Shanghai
  - Investigator site 0860052, Shanghai
  - Investigator site 0860042, Taiyuan
  - Investigator site 0860029, Wuhan
  - Investigator site 0860034, Wuhan
  - Investigator site 0860048, Xi'an
  - Investigator site 0860037, Xi'an
  - Investigator site 0860054, Xiangyang
- Investigator site 4200010, Hradec Králové, Czechia
- Denmark (3):
  - Investigator site 0450002, Aarhus
  - Investigator site 0450001, Copenhagen
  - Investigator site 0450003, Odense
- France (10):
  - Investigator site 0330034, Angers
  - Investigator site 0330013, Bordeaux
  - Investigator site 0330033, Clermont-Ferrand
  - Investigator site 0330025, Garches
  - Investigator site 0330023, Le Kremlin-Bicêtre
  - Investigator site 0330024, Limoges
  - Investigator site 0330022, Nantes
  - Investigator site 0330021, Nice
  - Investigator site 0330035, Paris
  - Investigator site 0330020, Strasbourg
- Georgia (5):
  - Investigator site 9950020, Kutaisi
  - Investigator site 9950005, Tbilisi
  - Investigator Site 9950002, Tbilisi
  - Investigator Site 9950003, Tbilisi
  - Investigator Site 9950004, Tbilisi
- Germany (11):
  - Investigator site 0490018, Berlin
  - Investigator site 0490017, Berlin
  - Investigator site 0490044, Bochum
  - Investigator site 0490013, Cologne
  - Investigator site 0490045, Essen
  - Investigator site 0490021, Göttingen
  - Investigator site 0490014, Hanover
  - Investigator site 0490016, Kiel
  - Investigator site 0490020, Leipzig
  - Investigator site 0490019, Potsdam
  - Investigator site 0490015, Regensburg
- Hungary (2):
  - Investigator site 0360017, Budapest
  - Investigator site 0360018, Kistarcsa
- Israel (3):
  - Investigator site 9720006, Holon
  - Investigator site 9720005, Ramat Gan
  - Investigator site 9720004, Tel Aviv
- Italy (11):
  - Investigator site 0390022, Brescia
  - Investigator site 0390029, Florence
  - Investigator site 0390024, Genova
  - Investigator site 0390027, Messina
  - Investigator site 0390003, Milan
  - Investigator site 0390026, Milan
  - Investigator site 0390007, Napoli
  - Investigator site 0390023, Pisa
  - Investigator site 0390008, Roma
  - Investigator site 0390028, Siena
  - Investigator site 0390042, Torino
- Japan (23):
  - Investigator site 0810035, Bunkyō City
  - Investigator site 0810002, Chiba
  - Investigator site 0810034, Chūōku
  - Investigator site 0810030, Fuchū
  - Investigator site 0810031, Fukuoka
  - Investigator site 0810065, Ginowan
  - Investigator site 0810066, Hakodate
  - Investigator site 0810058, Hiroshima
  - Investigator site 0810029, Kawaguchi
  - Investigator site 0810062, Kawasaki
  - Investigator site 0810026, Kodaira
  - Investigator site 0810061, Kyoto
  - Investigator site 0810027, Mibu
  - Investigator site 0810032, Nagoya
  - Investigator site 0810003, Osaka
  - Investigator site 0810007, Osaka
  - Investigator site 0810028, Sagamihara
  - Investigator site 0810033, Sapporo
  - Investigator site 0810037, Shinjuku-Ku
  - Investigator site 0810063, Suita
  - Investigator site 0810036, tabashi City
  - Investigator site 0810064, Tokushima
  - Investigator site 0810060, Yokohama
- Investigator site 3710001, Riga, Latvia
- Netherlands (2):
  - Investigator site 0310010, Amsterdam
  - Investigator site 0310011, Rotterdam
- Poland (7):
  - Investigator site 0480019, Bialystok
  - Investigator site 0480023, Katowice
  - Investigator site 0480017, Krakow
  - Investigator site 0480024, Krakow
  - Investigator site 0480020, Lodz
  - Investigator site 0480018, Lublin
  - Investigator site 0480022, Warsaw
- Romania (4):
  - Investigation site 0400002, Brasov
  - Investigator site 0400001, Bucharest
  - Investigator site 0400004, Constanța
  - Investigator site 0400003, Timișoara
- Russia (8):
  - Investigator site 0070017, Kazan'
  - Investigator site 0070023, Kazan'
  - Investigator site 0070016, Moscow
  - Investigator site 0070020, Moscow
  - Investigator site 0070018, Perm
  - Investigator site 0070019, Rostov-on-Don
  - Investigator site 0070014, Saint Petersburg
  - Investigator site 0070021, Saransk
- Serbia (3):
  - Investigator site 3810001, Belgrade
  - Investigator site 3810003, Belgrade
  - Investigator site 3810004, Kragujevac
- Spain (7):
  - Investigator site 0340020, Alicante
  - Investigator site 0340021, Badalona
  - Investigator site 0340038, Barcelona
  - Investigator site 0340019, Córdoba
  - Investigator site 0340017, Madrid
  - Investigator site 0340018, Madrid
  - Investigator site 0340016, Seville
- Taiwan (7):
  - Investigator site 8860014, Kaohsiung City
  - Investigator site 8860015, Taichung
  - Investigator site 8860013, Tainan
  - Investigator site 8860011, Taipei
  - Investigator site 8860012, Taipei
  - Investigator site 8860016, Taipei
  - Investigator site 8860017, Taoyuan District
- Turkey (Türkiye) (5):
  - Investigator site 0900025, Bursa
  - Investigator site 0900023, Istanbul
  - Investigator site 0900021, Izmir
  - Investigator site 0900022, Samsun
  - Investigator site 0900024, Sarıçam
- Ukraine (9):
  - Investigator site 3800012, Dnipro
  - Investigator site 3800014, Dnipro
  - Investigator site 3800010, Ivano-Frankivsk
  - Investigator site 3800015, Kharkiv
  - Investigator site 3800013, Kyiv
  - Investigator site 380008, Lutsk
  - Investigator site 380009, Vinnytsia
  - Investigator site 3800015, Vinnytsia
  - Investigator site 3800011, Zaporizhzhya
- United Kingdom (7):
  - Investigator site 0440017, Glasgow
  - Investigator site 0440015, Inverness
  - Investigator site 0440026, London
  - Investigator site 0440016, Oxford
  - Investigator site 0440018, Sheffield
  - Investigator site 0440019, Stoke-on-Trent
  - Investigator site 0440028, Tooting

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Allen JA, Lin J, Basta I, Dysgaard T, Eggers C, Guptill JT, Gwathmey KG, Hewamadduma C, Hofman E, Hussain YM, Kuwabara S, Le Masson G, Leypoldt F, Chang T, Lipowska M, Lowe M, Lauria G, Querol L, Simu MA, Suresh N, Tse A, Ulrichts P, Van Hoorick B, Yamasaki R, Lewis RA, van Doorn PA; ADHERE Study Group. Safety, tolerability, and efficacy of subcutaneous efgartigimod in patients with chronic inflammatory demyelinating polyradiculoneuropathy (ADHERE): a multicentre, randomised-withdrawal, double-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2024 Oct;23(10):1013-1024. doi: 10.1016/S1474-4422(24)00309-0. PMID 39304241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ARGX-113-1802 enrolled a broad and global (North America, Asia, Europe, and the rest of the world [ROW]) population of treatment-naïve participants and participants who were previously treated for CIDP (corticosteroids, IVIg, or SCIg) with confirmed, active disease and a wide range of disease severity.
  A total of 322 participants received efgartigimod PH20 SC in Stage A, and 221 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B.
Groups:
- Stage A: Efgartigimod PH20 SC: Participants receiving efgartigimod PH20 SC in Stage A
- Stage B: Efgartigimod PH20 SC: Participants who completed stage A and received efgartigimod PH20 SC in stage B
- Stage B: Placebo PH20 SC: Participants who completed stage A and received placebo PH20 SC in stage B
Period: Stage A
Arm/Group | Stage A: Efgartigimod PH20 SC | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Started | 322 | 0 (Stage B only) | 0 (There was no Placebo PH20 SC group in Stage A)
Completed | 221 | 0 (Stage B only) | 0 (There was no Placebo PH20 SC group in Stage A)
Not Completed | 101 | 0 | 0
Not completed — Lack of Efficacy | 8 | 0 | 0
Not completed — All events required for primary analysis achieved (rolled over to ARGX-1113-1902) | 22 | 0 | 0
Not completed — Adverse Event | 20 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lack of efficacy before end of Stage A | 28 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Prohibited medications | 2 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0
Not completed — Other | 5 | 0 | 0
Period: Stage B
Arm/Group | Stage A: Efgartigimod PH20 SC | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Started | 0 (Stage A only) | 111 | 110
Completed | 0 (Stage A only) | 64 | 74
Not Completed | 0 | 47 | 36
Not completed — All events required for primary analysis achieved (rolled over to ARGX-1113-1902) | 0 | 35 | 26
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Prohibited medications | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Sponsor decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 3
Not completed — Other | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: A total of 322 participants received efgartigimod PH20 SC in Stage A, and 221 of the 322 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B. Therefore, the total number of participants was 322, not 543 which was automatically calculated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage A: Efgartigimod PH20 SC | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC | Total
Number analyzed (Participants) | 322 | 111 | 110 | 543
Age, Categorical [Count of Participants; unit: Participants] — Population: A total of 322 participants were enrolled in Stage A. Of those 322, 221 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B.
  Participants
    Stage A: number analyzed (Participants) | 322 | 0 | 0 | 322
    Stage A: <=18 years | 0 | 0 | 0 | 0
    Stage A: Between 18 and 65 years | 247 | 0 | 0 | 247
    Stage A: >=65 years | 75 | 0 | 0 | 75
    Stage B: number analyzed (Participants) | 0 | 111 | 110 | 221
    Stage B: <=18 years | 0 | 0 | 0 | 0
    Stage B: Between 18 and 65 years | 0 | 86 | 88 | 174
    Stage B: >=65 years | 0 | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A total of 322 participants were enrolled in Stage A. Of those 322, 221 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B.
  years
    Stage A: number analyzed (Participants) | 322 | 0 | 0 | 322
    Stage A | 54.0 (13.92) |  |  | 54.0 (13.92)
    Stage B: number analyzed (Participants) | 0 | 111 | 110 | 221
    Stage B |  | 54.5 (13.18) | 51.3 (14.47) | 52.9 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 322 participants were enrolled in Stage A. Of those 322, 221 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B.
  Participants
    Stage A: number analyzed (Participants) | 322 | 0 | 0 | 322
    Stage A: Female | 114 |  |  | 114
    Stage A: Male | 208 |  |  | 208
    Stage B: number analyzed (Participants) | 0 | 111 | 110 | 221
    Stage B: Female |  | 38 | 41 | 79
    Stage B: Male |  | 73 | 69 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 322 participants were enrolled in Stage A. Of those 322, 221 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B.
  Participants
    Stage A: number analyzed (Participants) | 322 | 0 | 0 | 322
    Stage A: Hispanic or Latino | 23 |  |  | 23
    Stage A: Not Hispanic or Latino | 288 |  |  | 288
    Stage A: Unknown or Not Reported | 11 |  |  | 11
    Stage B: number analyzed (Participants) | 0 | 111 | 110 | 221
    Stage B: Hispanic or Latino |  | 9 | 4 | 13
    Stage B: Not Hispanic or Latino |  | 99 | 102 | 201
    Stage B: Unknown or Not Reported |  | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 322 participants were enrolled in Stage A. Of those 322, 221 participants were randomized in a 1:1 ratio to efgartigimod PH20 SC (N=111) or placebo (N=110) in Stage B.
  Participants
    Stage A: number analyzed (Participants) | 322 | 0 | 0 | 322
    Stage A: American Indian or Alaska Native | 0 |  |  | 0
    Stage A: Asian | 89 |  |  | 89
    Stage A: Native Hawaiian or Other Pacific Islander | 1 |  |  | 1
    Stage A: Black or African American | 4 |  |  | 4
    Stage A: White | 211 |  |  | 211
    Stage A: More than one race | 0 |  |  | 0
    Stage A: Unknown or Not Reported | 17 |  |  | 17
    Stage B: number analyzed (Participants) | 0 | 111 | 110 | 221
    Stage B: American Indian or Alaska Native |  | 0 | 0 | 0
    Stage B: Asian |  | 33 | 34 | 67
    Stage B: Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0
    Stage B: Black or African American |  | 1 | 1 | 2
    Stage B: White |  | 73 | 71 | 144
    Stage B: More than one race |  | 0 | 0 | 0
    Stage B: Unknown or Not Reported |  | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Stage A: Percentage of Participants With Confirmed Evidence of Clinical Improvement(ECI)
Time Frame: Up to 12 weeks during the open-label stage A
Population: SAF-A (Stage A safety analysis set): Participants who received at least 1 dose or part of a dose of efgartigimod PH20 SC in Stage A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 322
percentage of participants | 66.5 [61.0 to 71.6]

2. Primary Outcome: Stage B: Time to First Adjusted INCAT Deterioration Compared to Stage B Baseline
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: mITT (modified intent-to-treat) analysis set; Participants who were randomized in Stage B and who received at least 1 dose or part of a dose of IMP in Stage B.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
Days | NA [NA to NA] — Insufficient number of participants with events, less than 50% of the participants had clinically deteriorated. | 140.0 [75.0 to NA] — Insufficient number of participants with events to calculate the upper limit of the confidence interval.
Statistical Analysis 1: Comparison: Stage B: Efgartigimod PH20 SC vs Stage B: Placebo PH20 SC; Test type: Superiority; Hazard Ratio (HR) = 0.394, 95% CI 2-sided [0.253 to 0.614]

3. Secondary Outcome: Stage A: Time to Initial Confirmed Evidence of Clinical Improvement (ECI)
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 322
days
  25th percentile | 22 [22.0 to 23.0]
  50th percentile (median) | 43.0 [31.0 to 51.0]
  75th percentile | 71.0 [70.0 to 78.0]

4. Secondary Outcome: Stage A: Change From Stage A Baseline to Last Assessment in Stage A, in Adjusted INCAT Score
Description: Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) scores range from 0-10 with a score of 10 indicating the greatest degree of disability.
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 316
score on a scale | -0.9 (1.71)

5. Secondary Outcome: Stage A: Change From Stage A Baseline to Last Assessment in Stage A, in Medical Research Council (MRC) Sum Score
Description: The Medical Research Council (MRC) Sum scores range from 0 to 60 with a lower score indicating greater muscle weakness.
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 318
score on a scale | 3.8 (0.41)

6. Secondary Outcome: Stage A: Change From Stage A Baseline to Last Assessment in Stage A, in I-RODS Disability Scores
Description: The Inflammatory Rasch-built Overall Disability Scale (I-RODS) score ranges from 0-100, with lower scores indicating the greatest degree of disability.
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 320
score on a scale | 7.7 (15.48)

7. Secondary Outcome: Stage A: Change From Stage A Baseline to Last Assessment in Stage A, in TUG Score
Description: The Timed Up and Go (TUG) score is calculated as the number of seconds needed to complete a series of actions. The longer time needed to complete this test (expressed in seconds) indicates lower mobility.
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 288
seconds | -4.3 (0.83)

8. Secondary Outcome: Stage A: Change From Stage A Baseline to Last Assessment in Stage A, in Mean Grip Strength
Description: This is measured with a handheld device called a vigometer
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilopascal (kPa)
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 317
Kilopascal (kPa)
  dominant hand | 12.3 (18.68)
  nondominant hand | 11.2 (21.12)

9. Secondary Outcome: Stage A: Exposure Adjusted Occurrence of Treatment-emergent Adverse Events and Serious Adverse Events
Description: Treatment-emergent (serious) AEs expressed in number of events/100 PYFU (participant years of follow-up)
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Number; unit: Events/100 PYFU
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 322
Events/100 PYFU
  Exposure Adjusted Occurrence of Treatment-emergent Adverse Events | 1343.1
  Exposure Adjusted Occurrence of Treatment-emergent Serious Adverse Events | 51.2

10. Secondary Outcome: Stage A: Pre-dosing Efgartigimod Serum Concentrations Over Time
Time Frame: Up to 13 weeks during the open-label stage A (12 weeks + optional 1 additional week to confirm evidence of clinical improvement (ECI))
Population: The number analyzed in rows decreases due to participants withdrawing from the study and missing participant data. Week 13 was an optional additional week for the confirmation of the ECI. PK-A (Stage A PK analysis set): Participants from the SAF-A for whom at least 1 serum PK concentration during Stage A is available
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 298
ug/mL
  Week 1 | 14.9 (6.92)
  Week 2: number analyzed (Participants) | 285
  Week 2 | 19.6 (8.55)
  Week 3: number analyzed (Participants) | 263
  Week 3 | 19.7 (9.62)
  Week 4: number analyzed (Participants) | 250
  Week 4 | 18.9 (9.96)
  Week 5: number analyzed (Participants) | 141
  Week 5 | 18.4 (8.38)
  Week 6: number analyzed (Participants) | 116
  Week 6 | 19.2 (9.62)
  Week 7: number analyzed (Participants) | 105
  Week 7 | 17.3 (8.89)
  Week 8: number analyzed (Participants) | 82
  Week 8 | 18.8 (8.93)
  Week 9: number analyzed (Participants) | 70
  Week 9 | 17.8 (8.84)
  Week 10: number analyzed (Participants) | 51
  Week 10 | 17.3 (7.62)
  Week 11: number analyzed (Participants) | 41
  Week 11 | 20.1 (9.64)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 20.0 (6.89)
  Week 13: number analyzed (Participants) | 9
  Week 13 | 14.9 (7.24)

11. Secondary Outcome: Stage A: Percent Changes From Stage A Baseline of Serum IgG Levels Over Time
Time Frame: as for outcome 10
Population: The number analyzed in rows decreases due to participants advancing to stage B or withdrawing from the study and missing patient data. Week 13 was an optional additional week for the confirmation of the evidence of clinical improvement (ECI). PD-A (Stage A PD analysis set): Participants from the SAF-A for whom at least 1 serum PD concentration during Stage A is available.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 321
percent change
  Percent change from Baseline to Week 1: number analyzed (Participants) | 294
  Percent change from Baseline to Week 1 | -36.1 (0.58)
  Percent change from Baseline to Week 2: number analyzed (Participants) | 287
  Percent change from Baseline to Week 2 | -54.6 (0.80)
  Percent change from Baseline to Week 3: number analyzed (Participants) | 256
  Percent change from Baseline to Week 3 | -63.5 (0.71)
  Percent change from Baseline to Week 4: number analyzed (Participants) | 257
  Percent change from Baseline to Week 4 | -66.2 (0.89)
  Percent change from Baseline to Week 5: number analyzed (Participants) | 145
  Percent change from Baseline to Week 5 | -67.9 (0.74)
  Percent change from Baseline to Week 6: number analyzed (Participants) | 123
  Percent change from Baseline to Week 6 | -67.7 (1.42)
  Percent change from Baseline to Week 7: number analyzed (Participants) | 108
  Percent change from Baseline to Week 7 | -66.4 (1.96)
  Percent change from Baseline to Week 8: number analyzed (Participants) | 86
  Percent change from Baseline to Week 8 | -64.5 (4.28)
  Percent change from Baseline to Week 9: number analyzed (Participants) | 73
  Percent change from Baseline to Week 9 | -68.8 (1.17)
  Percent change from Baseline to Week 10: number analyzed (Participants) | 57
  Percent change from Baseline to Week 10 | -67.1 (1.90)
  Percent change from Baseline to Week 11: number analyzed (Participants) | 44
  Percent change from Baseline to Week 11 | -70.0 (1.41)
  Percent change from Baseline to Week 12: number analyzed (Participants) | 25
  Percent change from Baseline to Week 12 | -67.3 (4.44)
  Percent change from Baseline to Week 13: number analyzed (Participants) | 16
  Percent change from Baseline to Week 13 | -51.0 (10.00)

12. Secondary Outcome: Stage A: Number of Participants With Binding Antidrug Antibodies (ADA) Towards Efgartigimod or Antibodies (Ab) Against rHuPH20 and Neutralizing Antibodies (NAb) Against Efgartigimod and/or rHuPH20
Time Frame: Up to 12 weeks during the open-label stage A
Population: The number of participants analyzed is different since it is based on the number of evaluable participants for each drug. For Ab and NAb against rHuPH20 only 316 participants were evaluable, whereas for ADA and NAb towards efgartigimod 317 participants were evaluable. IMM-A (Stage A immunogenicity analysis set): Participants from the SAF-A for whom at least 1 ADA sample during Stage A is available
Measure: Count of Participants; unit: Participants
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 317
Participants
  ADA towards Efgartigimod incidence | 20
  Ab towards rHuPH20 incidence: number analyzed (Participants) | 316
  Ab towards rHuPH20 incidence | 45
  NAb against Efgartigimod incidence | 1
  NAb against rHuPH20 incidence: number analyzed (Participants) | 316
  NAb against rHuPH20 incidence | 0

13. Secondary Outcome: Stage A: Changes From Stage A Baseline to Last Assessment in Stage A, in EQ-5D-5L Visual Analog Scale (VAS) Over Time
Description: Scores range from 0-100 with 100 indicating the best health state. Therefore, positive changes indicate higher health-related quality of life reported by the patient.
Time Frame: Up to 12 weeks during the open-label stage A
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage A: Efgartigimod PH20 SC
Number analyzed (Participants) | 275
score on a scale | 10.7 (1.34)

14. Secondary Outcome: Stage B: Time to CIDP Disease Progression
Description: Time to chronic inflammatory demyelinating polyneuropathy (CIDP) disease progression is defined by the time from first dose of double-blind IMP to the first I-RODS score decrease ≥4 points compared to Stage B baseline using the centile metric.
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
days | NA [247.0 to NA] — The median (95% CI) time to CIDP Disease Progression could not be calculated because less than 50% of the participants showed CIDP Disease Progression in the efgartigimod PH20 SC group | 85 [50.0 to 253.0]

15. Secondary Outcome: Stage B: Number of Participants With Improved Functional Level Compared to Stage B Baseline
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
Participants | 50 | 40

16. Secondary Outcome: Stage B: Change From Stage B Baseline to Last Assessment in Stage B, in Adjusted INCAT Score
Description: as for outcome 4
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 109
score on a scale | 0.1 (1.08) | 0.9 (1.98)

17. Secondary Outcome: Stage B: Change From Stage B Baseline to Last Assessment in Stage B, in MRC Sum Score
Description: The Medical Research Council (MRC) Sum scores range from 0 to 60 with a lower score indicating greater muscle weakness.
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 109
score on a scale | -0.3 (0.43) | -3 (0.86)

18. Secondary Outcome: Stage B: Change From Stage B Baseline to Last Assessment in Stage B, in 24-item I-RODS Disability Score
Description: as for outcome 6
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 108
score on a scale | 0.8 (12.33) | -7.0 (19.10)

19. Secondary Outcome: Stage B: Change From Stage B Baseline to Last Assessment in Stage B, in TUG Score
Description: as for outcome 7
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 108 | 102
seconds | 0.8 (0.36) | 1.9 (0.60)

20. Secondary Outcome: Stage B: Change From Stage B Baseline to Last Assessment in Stage B, in Mean Grip Strength
Description: This is measured with a handheld device called a vigometer
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Measure: Mean (Standard Deviation); unit: Kilopascal (kPa)
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 109
Kilopascal (kPa)
  dominant hand | 2.1 (13.29) | -8.2 (20.69)
  nondominant hand | 2.0 (17.33) | -6.9 (21.30)

21. Secondary Outcome: Stage B: Time to 10% Decrease in the 24-item I-RODS
Description: as for outcome 6
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
days | NA [260.0 to NA] — The median (95% CI) time to 10% decrease in I-RODS could not be calculated because less than 50% of the participants showed 10% decrease in I-RODS in the efgartigimod PH2O SC group | 111 [84.0 to NA] — Could not be calculated

22. Secondary Outcome: Stage B: Exposure Adjusted Occurrence of Treatment-emergent Adverse Events and Serious Adverse Events
Description: Treatment-emergent (serious) AEs expressed in number of events/100 PYFU (participant years of follow-up)
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: SAF-B (Stage B safety analysis set): Participants from the SCR who received at least 1 dose or part of a dose of IMP in Stage B
Measure: Number; unit: Events/100 PYFU
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
Events/100 PYFU
  treatment-emergent adverse events | 347.6 | 510.9
  serious adverse events | 14.1 | 19.0

23. Secondary Outcome: Stage B: Pre-dosing Efgartigimod Serum Concentrations Over Time
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: The number analyzed in rows decreases due to participants completing the study, withdrawing from the study, and missing participant data. PK-B (Stage B PK analysis set): Participants from the SAF-B for whom at least 1 serum PK concentration during Stage B is available
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
ug/mL
  Week 4: number analyzed (Participants) | 97 | 97
  Week 4 | 18.4 (10.3) | 0.267 (0.365)
  Week 8: number analyzed (Participants) | 88 | 63
  Week 8 | 17.2 (9.11) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 12: number analyzed (Participants) | 73 | 49
  Week 12 | 18.1 (9.48) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 16: number analyzed (Participants) | 62 | 45
  Week 16 | 16.9 (9.03) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 20: number analyzed (Participants) | 57 | 39
  Week 20 | 16.8 (8.36) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 24: number analyzed (Participants) | 48 | 32
  Week 24 | 16.0 (7.89) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 28: number analyzed (Participants) | 43 | 28
  Week 28 | 18.5 (10.2) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 32: number analyzed (Participants) | 39 | 26
  Week 32 | 18.0 (9.50) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 36: number analyzed (Participants) | 36 | 22
  Week 36 | 17.9 (10.7) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 40: number analyzed (Participants) | 35 | 22
  Week 40 | 16.2 (8.20) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 44: number analyzed (Participants) | 31 | 17
  Week 44 | 18.1 (10.2) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)
  Week 48: number analyzed (Participants) | 27 | 13
  Week 48 | 16.3 (8.18) | NA (NA) — Data was below the limit of quantification (< 0.200 ug/mL)

24. Secondary Outcome: Stage B: Percent Changes of Serum IgG Levels Over Time
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: The number analyzed in rows decreases due to participants completing the study, withdrawing from the study, and missing participant data. PD-B (Stage B PD analysis set): Participants from the SAF-B for whom at least 1 serum PD concentration during Stage B is available
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 110
percent change
  Percent change from Baseline to Week 4: number analyzed (Participants) | 100 | 106
  Percent change from Baseline to Week 4 | -68.2 (1.14) | -36.7 (1.91)
  Percent change from Baseline to Week 8: number analyzed (Participants) | 91 | 64
  Percent change from Baseline to Week 8 | -68.2 (1.24) | -10.9 (2.41)
  Percent change from Baseline to Week 12: number analyzed (Participants) | 75 | 54
  Percent change from Baseline to Week 12 | -69.8 (1.09) | -7.1 (2.54)
  Percent change from Baseline to Week 16: number analyzed (Participants) | 66 | 48
  Percent change from Baseline to Week 16 | -67.4 (1.49) | -2.1 (3.09)
  Percent change from Baseline to Week 20: number analyzed (Participants) | 57 | 42
  Percent change from Baseline to Week 20 | -67.8 (1.30) | 2.0 (3.61)
  Percent change from Baseline to Week 24: number analyzed (Participants) | 51 | 34
  Percent change from Baseline to Week 24 | -67.2 (1.52) | 1.7 (4.22)
  Percent change from Baseline to Week 28: number analyzed (Participants) | 45 | 33
  Percent change from Baseline to Week 28 | -67.9 (1.42) | -2.3 (4.31)
  Percent change from Baseline to Week 32: number analyzed (Participants) | 38 | 27
  Percent change from Baseline to Week 32 | -68.5 (1.63) | 0.6 (5.18)
  Percent change from Baseline to Week 36: number analyzed (Participants) | 37 | 25
  Percent change from Baseline to Week 36 | -64.7 (2.82) | -3.6 (4.12)
  Percent change from Baseline to Week 40: number analyzed (Participants) | 36 | 23
  Percent change from Baseline to Week 40 | -68.0 (1.91) | -4.2 (4.98)
  Percent change from Baseline to Week 44: number analyzed (Participants) | 32 | 18
  Percent change from Baseline to Week 44 | -67.8 (1.92) | -3.6 (6.50)
  Percent change from Baseline to Week 48: number analyzed (Participants) | 31 | 17
  Percent change from Baseline to Week 48 | -66.6 (1.85) | -0.9 (7.36)

25. Secondary Outcome: Stage B: Number of Participants With Binding Antidrug Antibodies (ADA) Towards Efgartigimod or Antibodies (Ab) Against rHuPH20 and Neutralizing Antibodies (NAb) Against Efgartigimod and/or rHuPH20
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: IMM-B (Stage B immunogenicity analysis set): Participants from the SAF-B for whom at least 1 ADA sample during Stage B is available
Measure: Number; unit: participants
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 111 | 109
participants
  ADA towards Efgartigimod incidence | 2 | 64
  Ab towards rHuPH20 incidence | 52 | 32
  NAb against efgartigimod incidence | 0 | 13
  NAb against rHuPH20 incidence | 5 | 2

26. Secondary Outcome: Stage B: Changes From Stage B Baseline to Last Assessment in Stage B, in EQ-5D-5L Visual Analog Scale (VAS) Over Time
Description: as for outcome 13
Time Frame: Up to 48 weeks during the randomized placebo-controlled stage B
Population: as for outcome 22
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
Number analyzed (Participants) | 97 | 90
score on a scale | 0.5 (1.77) | -10.2 (2.47)

ADVERSE EVENTS:
Time Frame: 60 weeks (12 weeks during Stage A and 48 weeks during Stage B)
Description: Adverse events will be assessed at each participant visit. Treatment-emergent adverse events are reported in these tables.
Arm/Group | Stage A: Efgartigimod PH20 SC | Stage B: Efgartigimod PH20 SC | Stage B: Placebo PH20 SC
All-Cause Mortality (participants affected / at risk) | 2/322 | 0/111 | 1/110
Serious Adverse Events (participants affected / at risk) | 21/322 | 6/111 | 6/110
Other Adverse Events (participants affected / at risk) | 60/322 | 31/111 | 15/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage A: Efgartigimod PH20 SC (N=322) | Stage B: Efgartigimod PH20 SC (N=111) | Stage B: Placebo PH20 SC (N=110)
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 PNEUMONIA (Infections and infestations) | 1 | 1 | 0
SUSPECTED COVID-19 (Infections and infestations) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CHRONIC INFLAMMATORY DEMYELINATING POLYRADICULONEUROPATHY (Nervous system disorders) | 14 | 0 | 1
QUADRIPARESIS (Nervous system disorders) | 1 | 0 | 0
CALCULUS URINARY (Renal and urinary disorders) | 1 | 0 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 2
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 0 | 1 | 0
URINARY BLADDER POLYP (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage A: Efgartigimod PH20 SC (N=322) | Stage B: Efgartigimod PH20 SC (N=111) | Stage B: Placebo PH20 SC (N=110)
INJECTION SITE ERYTHEMA (General disorders) | 33 | 6 | 0
HEADACHE (Nervous system disorders) | 16 | 4 | 2
INJECTION SITE BRUISING (General disorders) | 4 | 6 | 1
COVID-19 (Infections and infestations) | 6 | 19 | 14
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 2 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04281472/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT04281472/SAP_001.pdf